CLINICAL TRIAL: NCT06346652
Title: Effects of Core Strengthening and PNF Pattern on Static Balance and Plantar Pressure in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Safa Saleem, Dr. Safa Saleem, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-216-03-2024
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Chronic Stroke
Keywords: core strengthening; plantar pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Routine Physical Therapy
  Interventions: Other: Routine Physical Therapy
- Interventional Group (Experimental): Routine Physical Therapy + PNF + Core Strengthening
  Interventions: Other: Routine Physical Therapy+ PNF and Core Stregthening

INTERVENTIONS:
Other: Routine Physical Therapy — Routine physical therapy involving muscle strengthening exercises, range of motion exercises and stretching exercises up to patient's tolerance. Other exercises were pelvic bridging, rolling, sitting and standing exercises, walking practice and balancing in parallel bars, wobble board exercises. Each session was of 60 minutes 5 times weekly for 6 weeks.
  Arms: Control Group
Other: Routine Physical Therapy+ PNF and Core Stregthening — Routine physical therapy for 20 minutes and additionally PNF technique (rhythmic initiation, and then agonistic reversals were performed in lower extremity in D1 flexion pattern and D1 extension pattern up to patient's tolerance and core strengthening for 20 minutes 5 times weekly for 6 weeks.
  Arms: Interventional Group

SUMMARY:
Stroke is a neurological disease characterized by neurological deficits caused by insufficiency of blood supply to brain. Disruption of blood supply to brain can be due to blockage of blood supply (ischemic) or leakage of blood in brain due to rupture of blood vessel (hemorrhagic). 90.5% of global occurrence of stroke was subjected to modifiable risk factors according to Global Burden of Disease study.

This study aims to compare the effects of core strengthening and proprioceptive neuromuscular facilitation on static standing balance and plantar pressure in chronic stroke patients.

DETAILED DESCRIPTION:
Background: Stroke is a neurological disease characterized by neurological deficits caused by insufficiency of blood supply to brain. Disruption of blood supply to brain can be due to blockage of blood supply (ischemic) or leakage of blood in brain due to rupture of blood vessel (hemorrhagic). 90.5% of global occurrence of stroke was subjected to modifiable risk factors according to Global Burden of Disease study.

Objective: To compare the effects of core strengthening and proprioceptive neuromuscular facilitation on static standing balance and plantar pressure in chronic stroke patients.

Methodology: 73 patients were enrolled in this study, 37 patients were assigned into control group while 36 participants were assigned into experimental group. Control group received routine physical therapy while experimental group received core strengthening and proprioceptive neuromuscular technique. Static component of berg balance scale and PoData Stabiliometeric plate was used for plantar pressure and measurement of balance respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age (45-60 years)
* Score of 9 or Higher on static component of berg balance scale
* Having score of equal or less than 2 on Modified Ashworth scale
* Having score of greater than or equal to 24 on Mini Mental State Examination.
* First ever episode of stroke
* Duration of stroke greater than 6 months
* Both genders

Exclusion Criteria:

* Concurrent orthopedic conditions that may hamper standing
* Relevant psychiatric disorders that may prevent from following instructions.
* Medical drugs that may influence intervention
* Conditions contraindicating physical activity
* Use of Cardiac pace maker.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Static Standing Balance | 6 weeks
  Measure using static component of berg balance scale. The items are scored from 0 to 4 with a score of 0 representing an inability to complete the task. Score of 4 representing independent item completion.

SECONDARY OUTCOMES:
Plantar Pressure | 6 weeks
  Foot plantar pressure is the pressure field that acts between the foot and support surface during static standing. PoData Stabiliometric plate was used to measure it. Normal value is 16.67% of the body weight on 5th metatarsal.

CONTACTS AND LOCATIONS:
Overall Officials: Safa Saleem, MSPTN, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No